CLINICAL TRIAL: NCT03536182
Title: CIPHER: A Prospective, Multi-Center Randomized Phase 3 Trial of Carbon Ion Versus Conventional Radiation Therapy for Locally Advanced, Unresectable Pancreatic Cancer
Brief Title: Trial of Carbon Ion Versus Photon Radiotherapy for Locally Advanced, Unresectable Pancreatic Cancer
Acronym: CIPHER
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to COVID and other recruitment issues the trial could not be initiated.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David Sher, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 022016-002
Record Dates: First submitted 2018-04-20; First posted 2018-05-24 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
Keywords: Pancreas; Adenocarcinoma.
MeSH Terms: conditions — Adenocarcinoma | interventions — Heavy Ion Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized in a 2:1 fashion (carbon:photon) between carbon ion radiotherapy or intensity modulated radiation therapy. Assuming a 10% dropout risk, the study will have 82% power to detect an increase in 2-year survival from 22% to 48% with carbon ion radiotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Arm A: Carbon ion radiotherapy (Active Comparator): The dose calculation algorithms used in Japan and Europe (local effect model, LEM) are different, so the total dose must be modified to ensure consistency
  1. Japan : 55.2 GyE in 4.6 GyE per fraction in 12 fractions delivered 4 days a week. At least 90% of each CTV receives at least 95% of the prescribed dose, and 100% of the GTV V95 must receive at least 95% of the prescribed dose.
  2. European: . Patients treated in Europe should receive 57.6 GyE in 4.8 GyE per fraction in 12 fractions delivered 4 days a week. At least 90% of CTV receives at least 95% of the prescribed dose, and 100% of the GTV V95 must receive at least 95% of the prescribed dose. This evaluation will occur in the LEM system
  Interventions: Radiation: Carbon Ion Radiation Therapy (CIRT)
- Arm B: Photon radiotherapy (Active Comparator): 50.4-56 Gy in 1.8-2.0 Gy per fraction in 28 fractions delivered 5 days a week. The plan should be normalized such that 100% of the PTV receives at least 48.9 Gy (i.e. 97% of 50.4 Gy). In addition, 100% of the GTV should receive at least 50.4 Gy. The maximum dose allowed to a point volume (0.03 mL) is 115% of the prescribed dose.
  Interventions: Radiation: Intensity Modulated Radiation Therapy (IMRT)

INTERVENTIONS:
Radiation: Carbon Ion Radiation Therapy (CIRT) — Patient will receive CIRT daily, 4 days a week for a total of 12 fractions/treatments plus concurrent chemotherapy (gemcitabine) weekly for 3 weeks. Gemcitabine will be given intravenously over about 1 hour in the outpatient clinic. Within 6 weeks of completing radiotherapy, patient will start 4 cycles of chemotherapy. If the doctor chooses gemcitabine+nab-Paclitaxel, patient will receive gemcitabine and nab-paclitaxel intravenously once a week for 3 weeks then 1 week off, for a total of 4 cycles (16 weeks). If the doctor chooses FOLFIRINOX, then patient will receive oxaliplatin, irinotecan, infusional 5-fluorouracil, and possibly leucovorin, all intravenously, every 2 weeks, for a total of 16 weeks.
  Arms: Arm A: Carbon ion radiotherapy
Radiation: Intensity Modulated Radiation Therapy (IMRT) — Patient will receive IMRT daily, 5 days a week for a total of 28 fractions/treatments plus concurrent chemotherapy (gemcitabine or capecitabine) weekly for 5 weeks. Gemcitabine will be given intravenously over about 1 hour in the outpatient clinic,within 6 weeks of completing radiotherapy,patient will start 4 cycles of chemotherapy. If the doctor chooses gemcitabine+nab-Paclitaxel, patient will receive gemcitabine and nab-paclitaxel intravenously once a week for 3 weeks then 1 week off, for a total of 4 cycles (16 weeks). If the doctor chooses FOLFIRINOX, then patient will receive oxaliplatin, irinotecan, infusional 5-fluorouracil, and possibly leucovorin, all intravenously, every 2 weeks, for a total of 16 weeks.
  Arms: Arm B: Photon radiotherapy

SUMMARY:
To determine if carbon ion radiotherapy improves overall survival versus photon therapy in patients with locally advanced, unresectable pancreatic cancer

DETAILED DESCRIPTION:
To compare the efficacy of carbon ion-based chemo radiotherapy with x-ray-based chemo radiotherapy for the treatment of locally advanced pancreatic adenocarcinoma by comparison of overall survival at 2 years following treatment.

Patient has 2 in 3 chance of receiving Arm A and 1 in 3 chance of receiving Arm B.

Arm A (chemoradiation takes place in Japan):

CIRT in 12 fractions/treatments plus concurrent gemcitabine, followed by 4 cycles of gemcitabine + nab-Paclitaxel, or until progression or intolerance of therapy

Arm B:

IMRT in 28 fractions plus concurrent gemcitabine or capecitabine, followed by 4 cycles of gemcitabine + nab-Paclitaxel, or until progression or intolerance of therapy

Per investigator discretion, patients may receive either:

1. Definitive treatment :
2. Neoadjuvant treatment:

Adjuvant chemotherapy 4 cycles of gemcitabine/nab-paclitaxel or FOLFIRNOX, Gemcitabine alone if these regimens are unavailable

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be willing and capable to provide informed consent within the 30 days prior to registration to participate in the protocol.
2. Histological and/or cytological diagnosis of pancreas adenocarcinoma must be done at any point prior to registration
3. Unresectable by radiographic or exploration within 30 days of registration
4. Age ≥ 18 years.
5. Distance from the pancreas tumor edge to the bowel and stomach > 3 mm (in both the prone and supine positions)
6. Tumor does not exceed 15 cm in greatest dimension
7. No evidence for metastatic disease as assessed by CT imaging of the chest, abdomen and pelvis OR by PET-CT within the 30 days prior to registration. Pancreas-protocol CT or magnetic resonance imaging (MRI) with gadolinium (for patients who cannot receive CT contrast) is required as part of this evaluation.
8. Zubrod performance status of 0-1, within 30 days prior to registration.
9. Adequate hematologic, renal, and liver function as defined by:Adequate hematologic, renal, and liver function as defined by:

   Absolute neutrophil count > 1500 cells/mm3 Creatinine <1.5 mg/dL Hemoglobin ≥ 8.0 g/dL AST and ALT < 2.5 X ULN Bilirubin ≤ 1.5 times the ULN (after stent placement, if necessary)
10. Patients must complete all required pretreatment evaluations
11. Able to travel to a foreign country within approximately 4 weeks of randomization (for patients enrolled outside of Japan and Italy)
12. If a patient receives 1 or 2 cycles of chemotherapy at an outside facility, pre-treatment laboratory values must meet the above criteria. If the protocol-compliant imaging had not been obtained prior to chemotherapy, they may be performed prior to registration and any additional chemotherapy being infused.
13. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

1. Subjects receiving other investigational agents.
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine or nab-paclitaxel or other agents used in study.
3. Subjects who are pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
4. Prior radiation to the upper abdomen
5. Placement of a metal stent for relief of biliary obstruction (metal stents may be placed following completion of radiation therapy).
6. Body weight >100 kg
7. Active inflammatory bowel disease or active gastric/duodenal ulcer
8. Metal implants in the upper abdomen
9. Expected medical intolerance of radiotherapy, concurrent chemotherapy, and/or adjuvant chemotherapy.
10. History of HIV or hepatitis B or C

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Over all Survival | 2 Years
  To compare the efficacy of carbon ion-based chemoradiotherapy with x-ray-based chemoradiotherapy for the treatment of locally advanced pancreatic adenocarcinoma by comparison of overall survival following treatment.

SECONDARY OUTCOMES:
Progression-free survival | 2 Years
  To compare progression-free survival between x-ray-based and carbon-ion-based chemoradiotherapy treatment courses for locally advanced pancreatic adenocarcinoma
Patterns-of-failure | 2 years
  To compare patterns-of-failure between x-ray-based and carbon-ion-based chemoradiotherapy treatment courses for locally advanced pancreatic adenocarcinoma
Quality-of-life Comparison | 12 Months
  To compare quality-of-life and toxicity outcomes between x-ray-based and carbon-ion-based chemoradiotherapy treatment courses for locally advanced pancreatic adenocarcinoma.The quality-of-life assessment will be performed during and after treatment. Patient-reported functional status will be assessed with the hepatobiliary subscales of the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep).
Toxicity using CTCAE 5.0 | 2 years
  Only adverse events assessed to be definitely, probably, or possibly related to protocol treatment will be considered. The rates of all Grade 3-5 adverse events, and death during or within 30 days of discontinuation of protocol treatment using CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: David Sher, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States
- National Institute of Radiological Sciences,4-9-1, Anagawa, Inage-ku,, Chiba, Japan